CLINICAL TRIAL: NCT01627366
Title: Survivorship Plans and Outcomes in Underserved Breast Cancer Survivors RCT
Brief Title: Study of Survivorship Care Plans and Outcomes in Underserved Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R01CA140481 (NIH)
Record Dates: First submitted 2012-06-04; First posted 2012-06-25 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2015-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Survivorship Care Plan (Experimental): Receipt of a personalized survivorship care plan and an in-person session with a trained nurse to review the contents of the care plan.
  Interventions: Other: Survivorship Care Plan
- Usual care (No Intervention): Receipt of usual medical care.

INTERVENTIONS:
Other: Survivorship Care Plan — Receipt of a personalized survivorship care plan and an in-person session with a trained nurse to review the contents of the care plan.
  Other Names: Treatment Summary and Survivorship Care Plans
  Arms: Survivorship Care Plan

SUMMARY:
Improvements in early detection and successful treatment of breast cancer have lead to a steady rise in the number of breast cancer (BC) survivors. With so many individuals living for extended periods after diagnosis, the Institute of Medicine (IOM) recommends the implementation of treatment summaries and survivorship care plans (TSSPs) as a mechanism to improve ongoing clinical and coordination of care, and to address the immediate post-treatment and long-term effects of cancer treatment, including the ongoing psychosocial burden of a cancer diagnosis. The need for TSSPs has also been strongly advocated by the American Society of Clinical Oncology's Quality Oncology Practice Initiative and TSSPs have been included in the recently introduced Comprehensive Cancer Improvement Act (H.R. 1844). This will be one of the first randomized controlled trials to test the efficacy of TSSPs.

The investigators will recruit 500 low income, medically underserved women from two county public hospitals, LAC+USC Medical Center and Harbor-UCLA Medical Center, 10-24 months after breast cancer diagnosis for participation in a randomized controlled trial (RCT) designed to test the efficacy of TSSPs. The investigators will randomize these women into one of two groups: 1) a control condition of usual medical care and 2) an experimental condition of the control condition + a tailored TSSP + 1 face-to-face nurse counseling session, with all cancer specialists and primary care physicians of record also receiving the TSSP and a cover letter suggesting how they can be clinically utilized.

The investigators specific aims are to assess and compare between experimental and control groups the following primary outcomes at one year post-intervention: 1) discussion and implementation of recommended breast cancer survivorship care, including surveillance and the evaluation and management of BC treatment-related symptoms, 2) patient satisfaction with survivorship communication and care, 3) pertinent aspects of health-related quality of life, and further, to then 4) assess the cost-consequences of the experimental intervention. This study will provide a unique opportunity to assess the efficacy of TSSPs in a low-income, underserved population of BC survivors known to be at high risk for poorer long-term outcomes, including in mental health, quality of life, recurrence and mortality, and will therefore allow us to demonstrate the greatest possible benefit of such an intervention.

DETAILED DESCRIPTION:
According to the National Cancer Institute (NCI), there are over 11 million cancer survivors in the United States. Among survivors, breast cancer (BC) is the most common, with BC survivors accounting for 23% (approximately 2.5 million). A 2006 report by the Institute of Medicine (IOM), From Cancer Patient to Cancer Survivor: Lost in Transition, provided a comprehensive assessment of the health needs of cancer survivors including a recommendation for the implementation of treatment summaries and survivorship care plans (TSSPs) to promote coordinated care for cancer survivors and to address the immediate post-treatment and long-term effects of cancer treatment including the ongoing psychosocial burden of a cancer diagnosis, as well as the potential for later sequelae of treatment. Because of the ever increasing number of BC survivors, the fact that 98% of patients with local stage and 84% of patients with regional stage survive for at least 5 years after diagnosis, and the multimodal nature of BC treatment, providing a mechanism that summarizes, monitors and coordinates BC follow-up care and treatment is essential. The use of TSSPs has also been strongly advocated by the American Society of Clinical Oncology's (ASCO) - Quality Oncology Practice Initiative and TSSPs have been included in the recently introduced Comprehensive Cancer Improvement Act of 2009 (H.R. 1844). Further, it is apparent that patients themselves strongly desire written follow-up plans after treatment is ended. The IOM recommended that research should be undertaken to evaluate the impact and costs of such plans. To our knowledge, however, no randomized controlled trials of TSSPs or evaluations of their cost-effectiveness have been conducted in a low-income, medically underserved population.

In the proposed study, we will recruit 500 low income, medically underserved women from two county public hospitals, Los Angeles County + University of Southern California Medical Center (LAC+USC Medical Center) and Harbor-UCLA Medical Center, 10-24 months after breast cancer diagnosis for participation in a randomized control trial (RCT) designed to test the efficacy of TSSPs. The intervention will be delivered after collection of pre-intervention (baseline) measures. We will consent and randomize these women into one of two groups: 1) a control condition of usual medical care and 2) an experimental condition of usual medical care + tailored materials which includes the TSSP + 1 face-to-face nurse counseling session, with all cancer specialist and primary care physicians of record also receiving the TSSP and a cover letter suggesting how it is to be clinically utilized. The study will provide a unique opportunity to assess the feasibility and clinical utility of a tailored treatment summary and survivorship care plan in a vulnerable population of BC survivors known to be at high risk for poorer long-term outcomes, including in mental health, quality of life, BC recurrence and mortality, and will therefore allow us to obtain the greatest possible effect size of such an intervention.

We will conduct a randomized controlled trial to test the efficacy of Treatment Summaries and Survivorship Care Plans and accompanying nurse counseling. The TSSP will consist of 4 sections: 1) the breast cancer treatment summary and 2) a cognitively appropriate survivorship care plan including recommendations for follow-up breast cancer care for both the patient and the physician, 3) a special section targeted towards the physician, and 4) a list of local and national patient resources.

Those women who consent to participate will have pre-intervention measures collected (i.e., the baseline interview) and will be randomized to either the usual care condition or the experimental condition. Individuals in the experimental group will participate in a face-to-face session with a trained, bilingual nurse to review the contents of the TSSP. Follow-up measures on all participants will be collected at 12-months after delivery of the intervention. We will evaluate receipt of recommended breast cancer survivorship care, patient self-efficacy and satisfaction with communication with providers, health related quality of life, and cost-effectiveness of the intervention. In addition, all participants in the control group will receive a written copy of their individualized TSSP at the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 21 years of age or older
* English- or Spanish-speaking
* Diagnosis of ductal carcinoma in situ (DCIS) or Stage I, II, or III BC for the first time
* 10-24 months post-diagnosis
* At least 1 month post-chemotherapy completion

Exclusion Criteria:

* Previous cancer except non-melanomatous skin cancers or in situ non-breast cancers
* Pregnant and lactating women
* Patients receiving parenteral anti-cancer therapy, except trastuzumab
* Clinically apparent cognitive or psychiatric impairment
* Participation in another research study
* Current treatment for another cancer
* Male
* Residing outside of Los Angeles County
* Too ill to participate

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2012-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Provider Adherence Score (PAS) | One year post-intervention
  Discussion and implementation of recommended breast cancer (BC) survivorship care, including surveillance and the evaluation and management of BC treatment-related symptoms, bone health, weight, vasomotor symptoms, mammography, clinical breast examinations, and depression, as well as discussion of the patient's primary BC-related concern.

SECONDARY OUTCOMES:
Patient satisfaction | One year post-intervention
  Patient satisfaction with survivorship communication and care.
Quality of life | One year post-intervention
  Health-related quality of life
Cost-consequence analysis | One year post-intervention
  Assess the immediate cost of the intervention itself, the downstream costs specifically related to health-care utilization from the survivorship care plan recommendations, and the resulting health benefits, in a cost consequence analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Rose C Maly, MD, MSPH, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States